CLINICAL TRIAL: NCT04188717
Title: Incidence, Risk Factors, Predictors and Survival for Neurological Complications After Liver Transplantation- A Retrospective Analysis
Brief Title: Incidence, Risk Factors, Predictors and Survival for Neurological Complications After Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS - Liver Transplant-2
Record Dates: First submitted 2019-11-28; First posted 2019-12-06 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: Liver Transplant; Complications; Neurologic Complication; Postoperative Complications
Keywords: liver transplantation; neurological complications; postoperative complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Liver transplantation is the definitive treatment in patients with chronic liver disease. Neurological complications (NC) occur commonly after liver transplantation. The investigators aim to evaluate the incidence, risk factors and predictors of neurological complications in both living donor and deceased donor transplantation done in the hospital. Between January 2011 to December 2016, 253 liver transplant recipients were recruited for this study. The investigators recorded the incidence of neurological complications, their median time of onset, their relationship with etiology of chronic liver disease, and the risk factors for the complications. The investigators also studied the relationship of neurological complications with duration of hospital and ICU stay, and survival. Using multivariate forward regression analysis , the investigators developed a scoring system for prediction of neurological complications in liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing liver transplant surgery
* 18-65 years

Exclusion Criteria:

* pregnant patients
* Acute Liver Failure, Acute on Chronic Liver Failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent liver transplant surgery for the specified time period were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Neurological complications | 90 days
  type of neurological complication
Mortality | 90 days
  mortality due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Karthik T Ponnappan, DM, Principal Investigator — ILBS